CLINICAL TRIAL: NCT05046145
Title: Effects of Non-invasive Neuromodulation on Food Desire, Chewing Pattern, Executive Functions and Biochemical Markers of Inflammation and Oxidative Stress
Brief Title: Effects of Non-invasive Neuromodulation on Food Desire, Chewing Pattern, Executive Functions and Oxidative Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Marta Maria da Silva Lira Batista, Principal Investigator, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCSONCRAVINGFOOD
Record Dates: First submitted 2021-08-13; First posted 2021-09-16 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Craving; Mastication Disorder; Memory Disorders; Executive Dysfunction; Transcranial Direct Current Stimulation; Inflammation; Oxidative Stress
Keywords: Craving; Executive Dysfunction; Oxidative Stress; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Memory Disorders; Inflammation | interventions — Speech Therapy; Mastication

STUDY DESIGN:
Intervention Model Description: The study will be a randomized, double-blind, parallel clinical trial. Participants will receive real tDCS or tDCS sham for 10 sessions during the treatment period. The interstice period of the total intervention will be 15 days (2 subsequent weeks, 10 working days, to apply the intervention). The probabilistic, simple randomized sample will consist of participants with randomized food cravings into two groups, there will be subdivision to receive or not neuromodulation, according to the flowchart.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not know what treatment they will receive. The outcomes assessor does not know treatment aplicado in participants sham or real).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS + speech therapy+ sham (Experimental): Participants will receive real tDCS and tDCS sham for 5 sessions during each treatment period. The interstice period of the total intervention will be 25 days, with 15 days of wash out between the two interventions. The probabilistic, simple randomized sample will consist of participants with food cravings randomized into two groups, according to the presence or absence of changes in eating behavior and within each group there will be subdivision to receive or not neuromodulation, according to the flowchart
  Interventions: Behavioral: speech therapy for chewing + real tDCS
- sham + tDCS + speech therapy (Experimental): Participants will receive real tDCS and tDCS sham for 5 sessions during each treatment period. The interstice period of the total intervention will be 25 days, with 15 days of wash out between the two interventions. The probabilistic, simple randomized sample will consist of participants with food cravings randomized into two groups, according to the presence or absence of changes in eating behavior and within each group there will be subdivision to receive or not neuromodulation, according to the flowchart
  Interventions: Behavioral: speech therapy for chewing + real tDCS

INTERVENTIONS:
Behavioral: speech therapy for chewing + real tDCS — participants will be instructed to chew their food correctly during the tDCS session, but the participant does not know if the tdcs is real or sham.
  Other Names: speech therapy for chewing + sham tDCS

SUMMARY:
From the change in self-regulation, memory is inhibited, allowing individuals to suppress or ignore unwanted or outdated associations and thus help to filter information relevant to dietary goals from irrelevant information. Provoking changes in neuroplasticity and cortical excitability contribute to the regulation of neural activity. Both could be modified by applying direct electrical current to the sensorimotor cortex, with polarity/current-dependent results, and their effect would last for hours after the end of stimulation. Transcranial Direct Current Stimulation (tDCS), translated into Portuguese as Estimulação Transcraniana por Corrente Contínua (ETCC) is a neuromodulating tool in which a low-intensity electrical current is applied to the scalp to modulate neuronal activity.

ELIGIBILITY:
Inclusion Criteria:

* being a health professional at the HU-UFPI (higher and technical levels);
* both sexes;
* Age between 20 and 59 years old.

Exclusion Criteria:

* Participants with communication disabilities (outbound or inbound);
* Type 1 and 2 diabetes
* low Body Mass Index (BMI; below 18.5),
* intracranial metal clip and/or prostheses;
* Abrupt change in weight (> 5 kg) in the last six months;
* the use will be excluded recreational use of psychoactive drugs,
* Being a smoker or using nicotine (tablet / absorbent),
* Having had significant recent trauma or traumatic brain injury,
* Present history of epilepsy,
* to be pregnant or under suspicion
* Missing teeth;
* Medical diagnosis of eating disorder or any psychiatric disorder,
* Having or having had cancer,
* Diagnosis of heart disease.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
change in desire to consume food. | pre-intervention.
  Questionnaires of Intense Food Desires - Trait (QDIC-T) validated for Brazilian Portuguese. The higher the score, the greater the amount of food craving presented.The QDIC-T scale is done on a 6-point scale with scores ranging from 39 to 214 points.
change in desire to consume food. | post-intervention (immediately after the end of study participation).
  Questionnaires of Intense Food Desires - Trait (QDIC-T) validated for Brazilian Portuguese. The higher the score, the greater the amount of food craving presented. The QDIC-T scale is done on a 6-point scale with scores ranging from 39 to 214 points.
change in the executive brain functions - working memory | pre-intervention.
  Trial Making Test (A and B). Assessments with single measurements (measurement of time, in seconds, to perform the test).
  the measurement unit for evaluating the outcome of these tests will be the amount of errors presented and the execution time (in seconds). The shorter the time and fewer errors, the better the result.
change in the executive brain functions - cognitive flexibility | post-intervention (immediately after the end of study participation).
  Stroop Tests. Assessments with single measurements (measurement of time, in seconds, to perform the test).
  the measurement unit for evaluating the outcome of these tests will be the amount of errors presented and the execution time (in seconds). The shorter the time and fewer errors, the better the result.

SECONDARY OUTCOMES:
change in the final value of inflammation scores | pre-intervention.
  inflammation markers (PCR in serum). The biochemical dosage of all elements will be in mg/L, higher values will represent a higher concentration, that is, a greater degree of inflammatory processes.
change in the final value of inflammation scores | post-intervention (immediately after the end of study participation).
  inflammation markers (PCR in serum). The biochemical dosage of all elements will be in mg/L, higher values will represent a higher concentration, that is, a greater degree of inflammatory processes.
change in the final value of antioxidant activity | pre-intervention.
  antioxidant activity (Catalase in erythrocytes). The biochemical dosage of all elements will be in mg/L, higher values will represent a higher concentration, that is, a greater degree of inflammatory processes.
change in the final value of antioxidant activity | post-intervention (immediately after the end of study participation).
  antioxidant activity (Catalase in erythrocytes). The biochemical dosage of all elements will be in mg/L, higher values will represent a higher concentration, that is, a greater degree of inflammatory processes.
change in desire to consume food. | pre-intervention.
  Questionnaires of Intense Food Desires - State (QDIC-E); validated for Brazilian Portuguese. QDIC-E is made up of a five-point scale, ranging from 15 to 75 points. The higher the score, the greater the amount of food craving presented.
change in desire to consume food. | post-intervention (immediately after the end of study participation).
  Questionnaires of Intense Food Desires - State (QDIC-E); validated for Brazilian.Portuguese. The higher the score, the greater the amount of food craving presented. QDIC-E is made up of a five-point scale, ranging from 15 to 75 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Do Piauí, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No
THERE IS PREDICTION THAT THERE WILL BE UNDERLYING RESEARCH BASED ON THE RESULTS FOUND.

REFERENCES:
- [Background] Ljubisavljevic M, Maxood K, Bjekic J, Oommen J, Nagelkerke N. Long-Term Effects of Repeated Prefrontal Cortex Transcranial Direct Current Stimulation (tDCS) on Food Craving in Normal and Overweight Young Adults. Brain Stimul. 2016 Nov-Dec;9(6):826-833. doi: 10.1016/j.brs.2016.07.002. Epub 2016 Jul 15. PMID 27498606
- [Background] Martin AA, Davidson TL, McCrory MA. Deficits in episodic memory are related to uncontrolled eating in a sample of healthy adults. Appetite. 2018 May 1;124:33-42. doi: 10.1016/j.appet.2017.05.011. Epub 2017 May 4. PMID 28479407
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Kane MJ, Engle RW. Working-memory capacity and the control of attention: the contributions of goal neglect, response competition, and task set to Stroop interference. J Exp Psychol Gen. 2003 Mar;132(1):47-70. doi: 10.1037/0096-3445.132.1.47. PMID 12656297
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Santos Ferreira I, Teixeira Costa B, Lima Ramos C, Lucena P, Thibaut A, Fregni F. Searching for the optimal tDCS target for motor rehabilitation. J Neuroeng Rehabil. 2019 Jul 17;16(1):90. doi: 10.1186/s12984-019-0561-5. PMID 31315679
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Diamond A. Executive functions. Handb Clin Neurol. 2020;173:225-240. doi: 10.1016/B978-0-444-64150-2.00020-4. PMID 32958176
- See also: Ljubisavljevic M, Maxood K, Bjekic J, Oommen J, Nagelkerke N. — https://pubmed.ncbi.nlm.nih.gov/27498606/
- See also: Martin AA, Davidson TL, McCrory MA — https://pubmed.ncbi.nlm.nih.gov/28479407/